CLINICAL TRIAL: NCT05615948
Title: An Open-Label Clinical Trial of Simultaneous Administration of Oral Aspirin and Ketamine as Adjunct to Oral Antidepressant Therapy in Treatment-Resistant Depression
Brief Title: Oral Aspirin + Ketamine as Adjunct to Oral Antidepressant Therapy for Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01-22-MMC
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Analgesia; Ketamine; Peripheral Nervous System Agents; Central Nervous System Depressants; Neurotransmitter Agents; Anti-Inflammatory Agents; Physiological Effects of Drugs; Sensory System Agents; Analgesics, Non-Narcotic; Anti-Inflammatory Agents, Non-Steroidal; Depressive Symptoms
Keywords: Maimonides Medical Center; Psychiatry; Ketamine; Aspirin; Antipyretics; Peripheral Nervous System Agents; Sensory System Agents; NMDA receptor antagonist; Anesthetics, Dissociative; Excitatory Amino Acid Antagonists; Excitatory Amino Acid Agents; Cyclooxygenase Inhibitors; Oral Medications for depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Agnosia; Depression | interventions — Ketamine; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Other): All individuals 18 years old or older who have Major Depressive Disorder and have failed to achieve response or remission to at least one proven antidepressant trial with minimum affective dose for a duration of at least 6 weeks.
  Interventions: Drug: VTS-K

INTERVENTIONS:
Drug: VTS-K — Proprietary oral formulation of 486mg aspirin and 80mg ketamine
  Other Names: Ketamine + Aspirin

SUMMARY:
The purpose of this study is to assess the effects of simultaneous administration of oral aspirin and oral ketamine as a therapeutic for those with Treatment Resistant Depression.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effect of simultaneous administration of oral aspirin and oral ketamine, formulated for partial release in the oral cavity and partially swallowed, as an adjunct to the oral antidepressant on depressive symptoms in patients suffering from Treatment Resistant Depression (TRD) in outpatient Psychiatric Clinic. Investigators will evaluate the effects of simultaneous administration of oral aspirin and oral ketamine, on depressive symptoms.

This is a prospective open-label, proof of concept clinical trial of simultaneous administration of proprietary formulations of oral aspirin and ketamine in medically stable adult patients with a diagnosis of Treatment Resistant Depression. All eligible participants will commit to three visits. The first two visits are in-person at the clinic for administration of oral ketamine and oral aspirin. Participants will be under observation for at least two hours. Study participant's vital signs will be monitored, periodically. The last visit will be conducted remotely.

Adult patients 18 years of age and older, with a diagnosis of TRD presenting to the psychiatric clinic will be screened for enrollment by study team.

:

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Treatment Resistant Depression with Montgomery-Asberg Depression Rating Scale score >22 upon presentation to the clinic
* Treatment Resistant Depression is defined as Major Depressive Disorder that does not cease after at least 6 week trial of another class of antidepressants
* Unipolar Depression

Exclusion Criteria:

* Adult patients with recent or current suicidal ideation with an intent to act, homicidal ideations with an intent to act
* History of Bipolar Disorder, Obsessive Compulsive Disorder, antisocial personality disorder, borderline personality disorder, and congestive cardiac failure
* Uncontrolled hypertension (BP >140 mm Hg systolic and/or >90 mm Hg diastolic on two separate readings at the time of screening) or on 2 medications for hypertension
* Patients with unstable vital signs (systolic blood pressure <90 or>160 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min),
* History of Gastrointestinal hemorrhage, renal and hepatic insufficiency
* Allergy to Ketamine or Aspirin
* Active Substance Abuse Disorder
* Active psychosis
* Active Peptic Ulcer Disease
* Lithium Therapy
* Swallowing difficulty
* Consumption of Aspirin or NSAID's within 6 hours of arrival to the site
* Previous participation in this study; a patient may not re-enroll in another study while in this study
* Pregnant or breastfeeding

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms on the Montgomery-Åsberg Depression Rating Scale (MADRS). | 7 Days
  Montgomery-Asberg Depression Rating Scale has a range from 0 to 60, where the lower score indicates the better health status. Change in mean total Montgomery Asberg Depression Rating Scale (MADRS) score from the baseline (pre-dose day 1 ) and on day 7

SECONDARY OUTCOMES:
A change in depressive symptoms on the Montgomery-Åsberg Depression Rating Scale (MADRS) from the baseline (pre-dose on day 1 and 4) and 2 hours post-medication administration | 4 Days
  Montgomery-Asberg Depression Rating Scale has a range from 0 to 60, where the lower score indicates the better health status. Change in mean total Montgomery-Asberg Depression Rating Scale prior to dose administration on Day 1 and Day 4 compared to 2 hours after dose administration for each day.
Clinician-Administered Dissociative States Scale (CADSS) | 4 Days
  Measurement of dissociative symptoms. Clinician Administered Dissociative States Scale (CADSS) comprises 23 subjective items, each on a 5 point scale, a "0" represents absence of any adverse events and "4" represents a severely bothersome side effect. A total score ranges from 0-92, a lower score indicates a better health status.
  :
Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) | 4 Days
  Overall side effects as measured by the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). SERSDA has 9 items, each graded on a five point scale, with "0" representing the absence of any adverse effects and "4" representing a severely bothersome side effect.
Maximal sedative effects using Modified Observer's Assessment of Alertness and Sedation ( MOAA/S) | 4 Days
  Modified Observer's Alertness/Sedation Scale ( MOAA/S) uses a 6 point scale. A "0" indicates failure to respond to painful stimulus, "5" represents fully alert. .

CONTACTS AND LOCATIONS:
Overall Officials: Deepan Singh, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Daly EJ, Trivedi MH, Janik A, Li H, Zhang Y, Li X, Lane R, Lim P, Duca AR, Hough D, Thase ME, Zajecka J, Winokur A, Divacka I, Fagiolini A, Cubala WJ, Bitter I, Blier P, Shelton RC, Molero P, Manji H, Drevets WC, Singh JB. Efficacy of Esketamine Nasal Spray Plus Oral Antidepressant Treatment for Relapse Prevention in Patients With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Sep 1;76(9):893-903. doi: 10.1001/jamapsychiatry.2019.1189. PMID 31166571
- [Background] Wajs E, Aluisio L, Holder R, Daly EJ, Lane R, Lim P, George JE, Morrison RL, Sanacora G, Young AH, Kasper S, Sulaiman AH, Li CT, Paik JW, Manji H, Hough D, Grunfeld J, Jeon HJ, Wilkinson ST, Drevets WC, Singh JB. Esketamine Nasal Spray Plus Oral Antidepressant in Patients With Treatment-Resistant Depression: Assessment of Long-Term Safety in a Phase 3, Open-Label Study (SUSTAIN-2). J Clin Psychiatry. 2020 Apr 28;81(3):19m12891. doi: 10.4088/JCP.19m12891. PMID 32316080
- [Background] Ochs-Ross R, Daly EJ, Zhang Y, Lane R, Lim P, Morrison RL, Hough D, Manji H, Drevets WC, Sanacora G, Steffens DC, Adler C, McShane R, Gaillard R, Wilkinson ST, Singh JB. Efficacy and Safety of Esketamine Nasal Spray Plus an Oral Antidepressant in Elderly Patients With Treatment-Resistant Depression-TRANSFORM-3. Am J Geriatr Psychiatry. 2020 Feb;28(2):121-141. doi: 10.1016/j.jagp.2019.10.008. Epub 2019 Oct 17. PMID 31734084
- [Background] Ketterer MW, Brymer J, Rhoads K, Kraft P, Lovallo WR. Is aspirin, as used for antithrombosis, an emotion-modulating agent? J Psychosom Res. 1996 Jan;40(1):53-8. doi: 10.1016/0022-3999(95)00524-2. PMID 8730644
- [Background] Mendlewicz J, Kriwin P, Oswald P, Souery D, Alboni S, Brunello N. Shortened onset of action of antidepressants in major depression using acetylsalicylic acid augmentation: a pilot open-label study. Int Clin Psychopharmacol. 2006 Jul;21(4):227-31. doi: 10.1097/00004850-200607000-00005. PMID 16687994
- [Background] Ng QX, Ramamoorthy K, Loke W, Lee MWL, Yeo WS, Lim DY, Sivalingam V. Clinical Role of Aspirin in Mood Disorders: A Systematic Review. Brain Sci. 2019 Oct 29;9(11):296. doi: 10.3390/brainsci9110296. PMID 31671812
- [Background] Marland S, Ellerton J, Andolfatto G, Strapazzon G, Thomassen O, Brandner B, Weatherall A, Paal P. Ketamine: use in anesthesia. CNS Neurosci Ther. 2013 Jun;19(6):381-9. doi: 10.1111/cns.12072. Epub 2013 Mar 22. PMID 23521979
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884